CLINICAL TRIAL: NCT01505985
Title: Effect of a Nutritional Intervention on Hip Fracture Surgery Recovery
Brief Title: Hip Fracture Surgery and Oral Nutritional Supplements
Acronym: HIATUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NES1026CLI
Record Dates: First submitted 2011-12-22; First posted 2012-01-09 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Hip Fracture
Keywords: Hip fracture; SPPB; Functional recovery
MeSH Terms: conditions — Hip Fractures | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialized Oral Nutritional Supplement (Experimental)
  Interventions: Dietary Supplement: Oral nutritional Supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral nutritional Supplement — Specialized nutritional supplement for seniors
  Arms: Specialized Oral Nutritional Supplement
Dietary Supplement: Placebo — placebo product with no specific nutrients
  Arms: Placebo

SUMMARY:
Senior hip fracture patients are the most vulnerable to malnutrition and protein deficiency. Low protein intake, like vitamin D deficiency, contribute to an increased risk for hip fracture. Notably, several clinical trials with protein supplementation in senior hip fracture patients resulted in fewer deaths, shorter hospital stay, and a higher likelihood of return to independent living. The proposal is to test the effect of an oral nutritional supplement (ONS) which has been designed to meet the specific nutrient needs of senior bone and muscle health. The hypothesis is that this ONS will improve functional recovery after hip fracture (as measured by Short Physical Performance Battery (SPPB)), improve quality of life, improve muscle mass, and- decrease falls and hospital re-admission after hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Age (70+);
* Had an acute hip fracture and surgical treatment
* Able to walk at least 3 meters without assistance of another person, with or without a walking aid other than a wheeled walker prior to hip fracture MMSE >=18 (proxy will be informed in addition if MMS-score ≤ 24)
* Able to perform the SPPB at baseline
* No prior hip fracture
* Patient (and/or his/her legal representatives/relatives) understands the study procedure, alternative treatments available and risks involved with the study, and voluntarily agrees to participate by giving his/her (or his/her legal representative's/relatives) written informed consent.

Exclusion Criteria:

* Baseline visit can not be performed between the second and tenth postoperative day.
* Milk protein allergy
* Patients with conservative treatment for hip fracture
* Serum calcium adjusted for albumin of > 2.6 mmol/L
* Pathologic fracture in the last year (except for fractures due to osteoporosis)
* Chemo therapy / Radiation /antihormonal therapy due to cancer in the last year
* Treatment which has an effect on calcium metabolism (e.g. PTH, calcitonin, chronic cortisone intake > 5mg/day in the last 12 months (except for inhalation and sporadic infiltration))
* Oral vitamin D intake of more than 1000 IU per day during the last 3 months before the study
* Unwilling to stop multi-vitamin, calcium supplementation, and vitamin D supplementation during the trial (maximal calcium supplement intake 250mg/d; no additional vitamin D supplementation). We will inform the treating physician that we initiated vitamin D supplementation as standard of care.
* Severe visual or hearing impairment
* Unwilling or unable to take study medication
* Diseases with a risk of recurrent falling (e.g. Parkinson's disease/syndrome, Hemiplegia after stroke, symptomatic stenosis of the spinal canal, polyneuropathy, epilepsy, recurring vertigo, recurring syncope) BMI ≥ 40
* Estimated creatinine clearance < 15 ml/min (estimated Creatinine Clearance cockcroft and Gault)
* Malabsorption syndrome (celiac diseases, inflammatory bowel disease, hepatic and/or pancreas dysfunction)
* Diseases that may enhance serum calcium: sarcoidosis, lymphoma, primary hyperparathyroidism
* Kidney stone in the last 10 years
* Patient heavily consumes alcohol containing products defined as greater than (>) 3 drinks (beer, wine, or distilled spirits) of alcoholic beverages per day.
* Patients who are planning a stay in a "sunny" location (e.g. winter sun resort) for more than one month during the trial
* Medication which has an effect on serum 25-hydroxyvitamin D level (e.g. certain anticonvulsants (e.g. Phenobarbital, Carbamazepin, Phenytoin) M. Paget (Ostitis deformans)
* Inflammatory arthritis (e.g. rheumatoid arthritis, reiter syndrome, psoriasis arthritis)
* Uncontrolled metabolic conditions, or psychiatric conditions that might make tolerance or evaluation of the feeding formula difficult
* Severe acute and/or chronic disease that makes the performance of the study assessments impossible (e.g. severe infection/sepsis, myocardial infarction, heart failure, respiratory failure or renal failure);
* Patient is taking peripherally acting anti-adiposity drugs (e.g. Xenical®, formoline L112®, (Acomplia®))
* Patients taking protein supplements (>15g per serving more than once a week) or are unwilling to stop any protein supplements during the trial Participation in a study in the last 6 month, except for studies without drug-application, or any influence of the study-medication can be excluded
* Patient is unlikely to adhere to the study procedures, to keep appointments, or is planning to relocate during the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | 6 months

SECONDARY OUTCOMES:
Nutritional status | 6 months
Quality of Life | 6 months
Muscle strength | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari,, MD, DrPH, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich,Dept. of Rheumatology and Institute of Physical Medicine,, Zurich, Switzerland